CLINICAL TRIAL: NCT04824404
Title: Integrated Intervention Combining CBT4CBT-Buprenorphine + Recovery Coach for Office-based Buprenorphine
Brief Title: CBT4CBT-Buprenorphine + Recovery Coach for Office-based Buprenorphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87691
Record Dates: First submitted 2021-03-19; First posted 2021-04-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment As Usual (TAU) (No Intervention): Participants in the standard of care condition will receive the standard treatment at the recovery program, which consists of weekly or bi-weekly visits (at the discretion of the provider) to the clinic to meet with their provider and provide a sample of blood.
- CBT4CBT-Buprenorphine + Recovery Coach (Experimental): This condition will consist of the CBT4CBT-Buprenorphine intervention alongside weekly coaching sessions from a recovery professional
  Interventions: Behavioral: CBT4CBT-Buprenorphine + Recovery Coach

INTERVENTIONS:
Behavioral: CBT4CBT-Buprenorphine + Recovery Coach — This condition will consist of the CBT4CBT-Buprenorphine intervention alongside weekly coaching sessions from a recovery professionalCBT4CBT-Buprenorphine is an 8-session (module) system for teaching a wide range of CBT skills (understanding and changing patterns of substance use; coping with craving; refusing offers of drugs and alcohol; problem-solving skills; identifying and changing thoughts about drugs and alcohol; and improving decision-making skills)
  Other Names: CBT4CBT+ Recovery Coach
  Arms: CBT4CBT-Buprenorphine + Recovery Coach

SUMMARY:
To conduct an 8-week pilot, randomized trial evaluating the feasibility, acceptability, and efficacy of an integrated intervention involving CBT4CBT-Buprenorphine + Recovery Coach in a population of 60 individuals who meet current DSM criteria for opioid use disorder and are receiving buprenorphine treatment in primary care.

DETAILED DESCRIPTION:
In this pilot study, 50 individuals with OUD on buprenorphine will be randomized to either 1) standard of care (N=25) or (2)CBT4CBT-Buprenorphine + Recovery Coach (N=250). This will be an 8-week trial.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years)
* having a DSM-V diagnosis of OUD
* sublingual buprenorphine/naloxone and/or buprenorphine
* having initiated maintenance treatment for OUD for at least 30 days before the screening
* self-report or toxicology screening positive for any substance within 30 days of screening;
* willing to accept a random assignment to either TAU/CBT4CBT-Buprenorphine + Recovery Coach;
* having adequate computer skills

Exclusion Criteria:

* having a severe medical or psychiatric disability that could impair their ability to perform study-related activities (determined by the clinician)
* being pregnant or breastfeeding;
* being unable to independently read and/or comprehend the consent form or other study materials
* being unable to read/speak English;
* having current suicidal ideation based on the Patient Health Questionnaire-9.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Change in drug use | 0-8 weeks
  Using saliva toxicology tests

SECONDARY OUTCOMES:
Retention to buprenorphine | 3 month follow up
  enrollment in and receiving buprenorphine and/or other effective medication treatment for OUD which will be verified by either report from the treatment clinic or electronic medical record
Change in drug use | 1 and 3 month follow up
  Using saliva toxicology tests

OTHER OUTCOMES:
Commission errors | 0-8 weeks
  This score indicates the number of times e client responded but no target was presented. A fast reaction time and high commission error rate points to difficulties with impulsivity.
Selective attention | 0-8 weeks
  This outcome will be measured by the Stroop Color and Word Test. This Stroop Test has three parts that generate simple and complex reaction times. Averaging the two complex reaction time scores from the Stroop Test generates a domain score for "reaction time."
Cognitive performance through Electroencephalogram | 0-8 weeks
  This outcome will be measured by alpha, the dominant frequency in the human scalp EEG of adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Recovery Clinic, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No